CLINICAL TRIAL: NCT00259896
Title: A Randomized, Open-label, Placebo-controlled, Repeat-dose Study to Assess the Pharmacokinetics and Pharmacodynamics of 5 Micrograms Exenatide Administered Subcutaneously Twice Daily for 7 Days in Healthy Normal Volunteers and in Subjects With Type 2 Diabetes Mellitus
Brief Title: In-patient Study in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLP105330
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-01

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: exenatide; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: exenatide

SUMMARY:
This study is a placebo-controlled study in both healthy normal subjects and patients with Type 2 Diabetes Mellitus to assess the levels of exenatide in the bloodstream when it is given for 7 days, and to assess the impact this medication has on various substances in the blood. Assessments include repeat blood sampling and monitoring of any side effects.

ELIGIBILITY:
Inclusion Criteria:

* have type 2 diabetes mellitus that has been diagnosed for at least three months
* must be taking either (1) no medication for their diabetes or (2) taking metformin, a sulfonylurea, or metformin and a sulfonylurea
* must be willing to wash-out of these medications for 14 days prior to the start of the study
* must have bloodwork that meets certain criteria (for example, total cholesterol < 240 mg/dL)

Exclusion Criteria:

* must not have any other major illness other than diabetes

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-10

PRIMARY OUTCOMES:
Pharmacodynamic measurements during 7 days of dosing.

SECONDARY OUTCOMES:
Pharmacokinetic measurements during 7 days of dosing.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline